CLINICAL TRIAL: NCT06741618
Title: MyPEEPS Mobile Plus
Brief Title: MyPEEPS Mobile Plus: A Multi-Level HIV Prevention Intervention for Young MSM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other); Callen-Lorde Community Health Center (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Rebecca Schnall, RN, MPH, PhD, Mary Dickey Lindsay Professor of Disease Prevention and Health Promotion, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAU8894; R01MD019181 (NIH)
Record Dates: First submitted 2024-12-15; First posted 2024-12-19 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: HIV/AIDS
Keywords: PrEP; care navigation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Participants randomized to the control arm will receive standard of care information regarding sexual and other behaviors that potentiate one's risk for HIV infection, receipt of a fact sheet about PrEP and PEP, referrals to the local PrEP clinic, and referrals for local sexually transmitted disease testing, and will have access to the MyPEEPS Mobile App during the study.
  Interventions: Behavioral: MyPEEPS Mobile
- Intervention (Experimental): Participants randomized to the intervention arm will have access to the MyPEEPS mobile application and Electronic peer PrEP navigation for the entire 12-month study period.
  Interventions: Behavioral: MyPEEPS Mobile; Behavioral: Electronic PrEP peer navigation

INTERVENTIONS:
Behavioral: MyPEEPS Mobile — An evidence-based, digitally delivered mHealth sexual risk reduction intervention on HIV incidence
Behavioral: Electronic PrEP peer navigation — Electronic peer navigation to PreP services
  Arms: Intervention

SUMMARY:
MyPEEPS Mobile Plus, a multi-level intervention for improving HIV prevention outcomes in YMSM, is a novel and evidence-driven approach using mobile technology to deliver HIV prevention information specifically developed for YMSM. Building on strong preliminary work, the proposed research is the next logical step in a body of work designed to assess whether refinement of this mobile intervention used in combination with virtual PrEP Peer Navigation will result in improvements in PrEP uptake and a reduction in HIV-related behavior. This is key to advancing HIV prevention among HIV-negative US persons at extremely high-risk for HIV seroconversion.

DETAILED DESCRIPTION:
This study expands MyPEEPS Mobile to develop MyPEEPS Mobile Plus, a multi-level intervention comprised of MyPEEPS Mobile with added PrEP content (based upon expert advisory and youth feedback) + PrEP E-Peer Navigation to overcome the challenges of PrEP initiation, adherence, and persistence among YMSM. Peer navigation is an evidence-based, widely recommended intervention for reaching youth and MSM for HIV-related care outcomes, with evidence of acceptability among racial/ethnic minority YMSM for PrEP. Peer navigation addresses common reasons for failing to begin or maintain PrEP use, including low perceived risk, structural or logistic barriers to care engagement, and anticipated side effects. Relative to in-person and group-based HIV prevention programs, behavioral interventions with digital and virtual components can have vast reach and present unique potential to rapidly scale delivery to very large and hidden groups. Therefore, the investigators propose to conduct a randomized controlled trial to test the efficacy of MyPEEPS Mobile Plus (a multi-level intervention comprised of MyPEEPS Mobile + PrEP E-Peer Navigation) for promoting initiation, adherence, and persistence of PrEP and decreased HIV risk behavior in YMSM. Building upon the team's demonstrated ability to enroll large numbers of young racially and ethnically diverse YMSM and extensive experience developing mobile health interventions, the proposed study will test the efficacy of this expanded, multi-level mobile HIV prevention intervention emphasizing PrEP. If efficacious, it will increase PrEP initiation, adherence, and persistence and decrease overall HIV risk in diverse YMSM in the US.

ELIGIBILITY:
Inclusion Criteria:

* 16-25 years of age
* identify as male, non-binary, or genderqueer
* male sex assigned at birth
* understand and read English
* own a smartphone
* report condomless anal sex with a male in the past year
* HIV-negative (OraQuick verified)

Exclusion Criteria:

* HIV Positive
* If study staff determine participant unable to consent due to obvious and severe cognitive impairment or under the influence of drugs or alcohol
* Transgender identity
* currently report consistent use of PrEP

Ages: 16 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — male, nonbinary, genderqueer
Enrollment: 500 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
PrEP Initiation: | Baseline, 6-month follow-up, 12-month follow-up
  Participants will self-report attending at least one PrEP-related care visit to asess medical eligibility for PrEP initiation.

SECONDARY OUTCOMES:
PrEP Adherence | Baseline, 6-month follow-up, 12-month follow-up
  Daily oral PrEP users will report PrEP use in the past 7-days.
PrEP Persistence | Baseline, 6-month follow-up, 12-month follow-up
  Questions will be measure visit constancy, i.e., self-report at least 1 PrEP related care visit in the past 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Garofalo, MD, MPH, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago; Lisa Kuhns, PhD, MPH, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Columbia University, New York, New York, United States